CLINICAL TRIAL: NCT03107468
Title: The Effectiveness and Safety of Traditional Korean Medicine for Symptomatic Lumbar Spinal Spondylolisthesis: a Randomized Controlled International Collaborative Multi-center Trial
Brief Title: Korean Medicine for Symptomatic Lumbar Spinal Spondylolisthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kim Ki Ok (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Mayo Clinic (Other); Kyunghee University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Kim Ki Ok, President, Mokhuri Oriental Hospital
Organization: Mokhuri Oriental Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHNBH-16031
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Spondylolisthesis, Lumbosacral Region
Keywords: Non-surgical treatment; Acupuncture; Chuna; Physiotherapy; Epidural steroid injection
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent outcome assessors who do not know allocation result will participate in the outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mokhuri intensive treatment group (Experimental): Patients in this arm will be treated with 35-week of Mokhuri intensive treatment program which compromise 10 sessions of acupuncture, Chuna and patient consultation during 5 weeks.
  Interventions: Other: Mokhuri intensive treatment
- Non-surgical conventional treatment group (Active Comparator): Patients in this arm will be treated with 10 sessions of non-surgical conventional standard treatment including conventional drug treatment and injection treatment during 5 weeks.
  Interventions: Other: Non-surgical conventional standard treatment

INTERVENTIONS:
Other: Mokhuri intensive treatment — Patients in this arm will be treated with acupuncture, Chuna and patient consultation during 5 weeks. For acupuncture therapy, disposable sterile needles will be placed on LI4, ST36, LV3, B22, B23, B24 and B25 of both sides of a patient for 15 minutes. For Chuna therapy, the patient lies on the Ergo Style™ FX-5820 Table in the prone position and back muscles will be relaxed by manual manipulation during flexion and extension movement of the table for 5 to 6 minutes. Patient consultation regarding the precautions for everyday life, the precautions for activity in bed, the precautions for walking, the precautions for particular movements and the exercises will be offered for 5 minutes.
  Arms: Mokhuri intensive treatment group
Other: Non-surgical conventional standard treatment — Patients in this arm will be treated with 10 sessions of non-surgical conventional standard treatment including conventional drug treatment and injection treatment under the consultation of neurosurgeons or doctors of anesthesiology or rehabilitation medicine during 5 weeks. For drug therapy, muscle relaxants, NSAIDs, gabapentin, pregabalin or tricyclic antidepressants will be prescribe. For epidural steroid injection, 3cc of epidurals will be injected at the affected lesion once or twice. For physical therapy, participants shall participate in conventional physical therapy with the aid of physical therapists, including heating pad, deep tissue heating device and transcutaneous electrical nerve stimulation (TENS) twice a week during the five weeks of participation.
  Arms: Non-surgical conventional treatment group

SUMMARY:
This is a clinical trial for evaluating the safety and effectiveness of the Mokhuri intensive treatment program regarding pain and function before and after treatment between a group receiving the Mokhuri intensive treatment program (Chuna, acupuncture, and patient education) for five weeks and another group receiving non-surgical conventional standard treatment (drugs for pain relief, epidural steroid injection treatment, and physical therapy).

The trial will be conducted through international cooperation between Mayo Clinic in the United States and Mokhuri Oriental Medicine Hospital in Korea. All subjects in Korea and the US will be selected based on the same inclusion criteria and exclusion criteria. All subjects in the treatment arm will receive the same treatment in Korea and the US. In collaboration and with the support of Mayo Clinic's Department of Integrative Medicine and Health, and to ensure treatment consistency between Korea and the US, an acupuncturist from the USA will travel to Korea and train on-site for one month in Mokhuri hospital.

The trial subjects who agree to participate in the clinical trial after providing informed consent will receive the required examinations and tests according to the clinical trial plan. If they are appropriate for this clinical trial and eligible based on the Inclusion and exclusion criteria, they will be randomly assigned to the group that will undergo the focused Mokhuri intensive treatment program and to the group that will receive non-surgical conventional treatment on their second visit. All the subjects in this study will be educated regarding the study procedure and scheduled visits and will participate in the allocated treatments for five weeks. Afterwards, clinical outcomes of both groups will be evaluated after end of the treatments from between a week and five weeks (within +7 days). The clinical trial ends after the follow-up evaluations that will take place 12 weeks, 24 weeks, 48 weeks, and 96 weeks after the end of the treatment evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with all the following requirements will be included as appropriate subjects in the clinical trial:

  1. Those aged from 19 to 78 years
  2. Those with a diagnosis of degenerative lumbar spinal spondylolisthesis and have low back pain, lower limb radiating pain, or leg discomfort when standing or walking with severity of at least 50 in a 0 to 100 VAS for each symptom
  3. Those suffering from neurologic claudication or radicular pain at least for one year
  4. Those with neurogenic claudication within five minutes when walking on a treadmill at the speed of 1.5 miles per hour
  5. Those not receiving epidural injection treatments within the past one month
  6. Those who have not undergone lumbar surgery
  7. Those who confirmed spondylolisthesis on L-spine AP, lateral & both oblique views
  8. Those who weigh 250 lbs (113.398 kg) or less
  9. Those who are 2.1 m (6.890 ft) in height or shorter
  10. Those agreeing to participate in this clinical trial after receiving a thorough explanation of the purposes and characteristics of the trial and who have also signed the written informed consent form.

Exclusion Criteria:

* Subjects will be excluded for the following conditions:

  1. Those with a history of diseases in the past or in the present that cause ambulatory functional disability
  2. Those with knee joint and hip joint disorders that severely limit walking (i.e. moderate or severe osteoarthritis in the knee or hip joints)
  3. Those who has been diagnosed as peripheral blood vessel diseases or vascular diseases in the past, shows an ankle-brachial index (ABI) below 0.9 or is diagnosed as peripheral artery disease by Doppler ultrasonography of lower limbs, if necessary
  4. Those with severe diseases (cardiac disorders or renal insufficiency) such that the ambulatory evaluation is not attainable
  5. Those with other specific spinal diseases (ankylosing spondylitis, spinal osteomyelitis, metabolic diseases, severe osteoporosis, etc.)
  6. Those with severe neurological defects including foot drop or cauda equina syndrome
  7. Those with spinal instability confirmed by L-spine x-ray flexion and extension views. Spinal instability will be defined as observing one or more of the following: 4.5 mm sagittal plane translation, 20 degrees of sagittal plane rotation at L4-5, or 25 degrees of sagittal plane rotation at L5-S1.
  8. Those with malignancy
  9. Those with psychiatric conditions such as major depressive disorder and anxiety disorder in the past or present (e.g., panic disorder, episodes of mania, delusion, and schizophrenia)
  10. Those using narcotic analgesics, including the external dosage form or patch
  11. Those on medications for respiratory diseases including gastritis, stomach ulcer, and irritable bowel syndrome
  12. Pregnant women, lactating women, or those planning to become pregnant
  13. Those who appear likely to encounter difficulties in adhering to this protocol such as those regarding treatment, hospitalization, or preparation for the survey
  14. Those subjects who the clinical investigators judge to be inappropriate

Ages: 19 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
0 to 100 Visual Analogue Scale (VAS) for low back pain | 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 18th, 30th, 54th and 102th weeks
  The degree of pain recognized as backache is indicated on a 100 mm straight line. The participant is to indicate the average level of lumbar pain experienced for the past one week.

SECONDARY OUTCOMES:
0 to 100 Visual Analogue Scale (VAS) for leg pain | 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 18th, 30th, 54th and 102th weeks
  The degree of pain recognized as leg pain is indicated on a 100 mm straight line. The participant is to indicate the average level of lumbar pain experienced for the past one week.
EQ-5D | 2nd, 3rd, 4th, 5th, 6th, 7th, 18th, 30th, 54th and 102th weeks
  For assessing quality of life, participants must place checkmarks at the most appropriate points in response to inquiries on each of the five items regarding their health conditions.
Oswestry Disability Index | 2nd, 3rd, 4th, 5th, 6th, 7th, 18th, 30th, 54th and 102th weeks
  ODI is the index derived from the Oswestry disability questionnaire (ODQ) for assessing the degree of pain, sleep disturbance, self-treatment, walking, sitting, standing, moving, sexual life, social activities, and travel.
Roland-Morris Disability Questionnaire (RMDQ) | 2nd, 6th, 7th, 18th, 30th, 54th and 102th weeks
  The Roland-Morris Disability Questionnaire (RMDQ) is a tool that is widely used for evaluating the functional conditions of patients with low back pain.
Zurich Claudication Questionnaire (ZCQ) | 2nd, 6th, 7th, 18th, 30th, 54th and 102th weeks
  Zurich Claudication Questionnaire (ZCQ) is an instrument for assessing pain and symptoms related to the spinal stenosis.
Walking duration and distance free of leg pain | 2nd, 3rd, 4th, 5th, 6th, 7th, 18th, 30th, 54th and 102th weeks
  Patients walk on the revolving tracks to a distance of 25m at their preferred speed.
The ratio between the actual duration of participation and the originally scheduled duration in each group | 7th week
  Participants whose 0 to 100 VAS for back pain and leg pain would decrease below 10 at every-week evaluation will stop the treatment immediately. The numbers of patients who stop the scheduled treatments early and finished full scheduled treatments will be assessed in each group and the differences in the ratio between groups will be assessed.
Treadmill test | 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 18th, 30th, 54th and 102th weeks
  The patients shall walk on the level treadmill at a speed of 1.5 miles (2.414 km/sec). The time until they feel pain in their legs is to be measured.
Adverse event assessments | 2nd, 3rd, 4th, 5th, 6th, 7th, 18th, 30th, 54th and 102th weeks
  . Participants voluntarily report adverse events and experiments are needed to observe them on a regular basis.
Investigation for the presence of any additional spondylolisthesis treatment and the types thereof | 18th, 30th, 54th and 102th weeks
  Concomitant medication or treatments will be recorded during the follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Kiok Kim, Dr., Principal Investigator — Mokhuri Oriental Medicine Hospital
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Mokhuri Oriental Medicine Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim K, Yan D, Bauer BA, Choi JC, Wang Z, Jung JE, Kim J, Kim TH, Eldrige JS, Mauck WD, Holmes BD, Bublitz SE, Seo M, Qu W. Nonsurgical Integrative Treatments for Symptomatic Degenerative Lumbar Spondylolisthesis: A Multinational Randomized Controlled Clinical Trial. Mayo Clin Proc. 2025 Nov 2:S0025-6196(25)00334-9. doi: 10.1016/j.mayocp.2025.05.030. Online ahead of print. PMID 41176728
- [Derived] Kim K, Youn Y, Lee SH, Choi JC, Jung JE, Kim J, Qu W, Eldrige J, Kim TH. The effectiveness and safety of nonsurgical integrative interventions for symptomatic lumbar spinal spondylolisthesis: A randomized controlled multinational, multicenter trial protocol. Medicine (Baltimore). 2018 May;97(19):e0667. doi: 10.1097/MD.0000000000010667. PMID 29742708